CLINICAL TRIAL: NCT07229690
Title: Appendicular Stump Closure Techniques
Brief Title: Closure of Appendicular Stump
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, prof, Zagazig University
Other Study IDs: appendicular stump closure
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Appendix
Keywords: appendix; stump

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- endoloop: closure of stump by endoloop
  Interventions: Procedure: endoloop closure
- intracorporeal suture: closure of stump by suture
  Interventions: Procedure: intracorporeal suture

INTERVENTIONS:
Procedure: endoloop closure — closure of stump by endoloop
  Groups: endoloop
Procedure: intracorporeal suture — closure of stump by suture
  Groups: intracorporeal suture

SUMMARY:
this study compare between different types of appendicular stump closure

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years a clinical diagnosis of complicated AA

Exclusion Criteria:

* • Pregnancy (n=7)

  * Complicated appendicitis secondary to colon caecum (n=2)
  * inflammatory bowel disease (n=4)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with complicated acute appendicitis
Sampling Method: Probability Sample
Enrollment: 666 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
appendicular leak | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Tamer.A.A.M. Habeeb, Principal Investigator — Zagazig University
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes